CLINICAL TRIAL: NCT00999193
Title: Effectiveness and Cost-effectiveness of Conservative and Operative Treatment of Three- and Four-part Fractures of the Proximal Humerus. A Nested Randomised Controlled Trial and Cohort Study
Brief Title: Proximal Humeral Comminuted Fractures in the Elderly - PERCELE Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment decline and research question getting outdated
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Tuomas Lahdeoja, MD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS-428/13/03/02/08
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Humeral Fracture
Keywords: Shoulder; Fracture; Locking Plate; Hemiarthroplasty; Conservative; Comminuted Proximal Humerus Fracture
MeSH Terms: conditions — Humeral Fractures; Fractures, Bone | interventions — Hemiarthroplasty; Conservative Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conservative Treatment (Active Comparator)
  Interventions: Other: Conservative treatment
- ORIF w. locking plate, no luxation (Experimental)
  Interventions: Procedure: locking plate, ORIF
- Hemiarthroplasty, no luxation (Experimental)
  Interventions: Procedure: Hemiarthroplasty

INTERVENTIONS:
Procedure: locking plate, ORIF — Open reduction of the fracture (and GH joint), internal fixation with a locking plate. Tuberculum fragments are sutured to the plate with thick non-absorbable suture.
  Arms: ORIF w. locking plate, no luxation
Procedure: Hemiarthroplasty — Replacement of the humeral articular head with hemiprosthesis. Tubercles are sutured to the prosthesis with thick nonabsorbable sutures.
  Arms: Hemiarthroplasty, no luxation
Other: Conservative treatment — Immobilisation in a supporting brace for 3 weeks, then increasingly active rehabilitation program supported by a physiotherapist until 12 weeks of the injury.
  Arms: Conservative Treatment

SUMMARY:
Fractures of the proximal humerus are common in elderly patients. The optimal treatment of comminuted, displaced fractures is subject to controversy, and the results of operative treatment have not been shown to be superior to conservative treatment. The aim of the study is to compare locking plate osteosynthesis versus treatment with fracture hemiarthroplasty versus conservative treatment in a randomised, controlled protocol. The results of treatment are measured at 6 weeks, 3 months, 6 months, 12 months and 24 months. Main outcome measures are Pain at rest and activity (NRSs) and functional assessment of the shoulder with Constant Score. Secondary outcome measures are Simple Shoulder test (SST), Disabilities of the Arm, Shoulder and Hand (DASH), quality of life assessment (15D), subjective patient satisfaction and costs. The study also has a cohort follow-up of the patiens who decline randomisation.

The recruitment target was 90 patients, but the study recruitment was stopped due to slow recruitment (too few patients presenting with eligibile injury to the hospital) at 60 patients in November 2019.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Acute trauma: 1. randomisation (op vs cons) within 7 days of injury.
* 3- or 4-part fracture with >5mm dislocation of the anatomic neck.

  * AO classification C1-2 for non-luxation fractures
  * AO classification C3 for luxation fractures

Exclusion Criteria:

* Head Splitting fracture
* Open fracture
* Additional fractures in the shoulder region
* Other injuries requiring surgical treatment
* Clinically significant injury of the brachial plexus or vasculature
* Pathological fracture associated with cancer
* History of a fracture of the clavicle, scapula or humerus, or history of a very significant disease or trauma of the shoulder region (hemiparesis, tumour, osteomyelitis, grave arthrosis etc)
* Rheumatoid Arthritis in the shoulder requiring active treatment
* Reduced co-operation or incapability for independent living (dementia, mental illness, drug- or alcohol abuse etc)
* unwillingness to accept some of the treatment options.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Pain at rest Numeric Rating Scale 0-10 (NRS) | 6 weeks, 3 mo, 6 mo, 1 year, 2 years
Pain in active motion NRS | 6 weeks, 3 mo, 6 mo, 1 year, 2 years
Constant Score | 3 mo, 6 mo, 1 year, 2 years

SECONDARY OUTCOMES:
Simple Shoulder Test (SST) | 3 mo, 6 mo, 1 year, 2 years
Disabilities of the Arm, Shoulder and Hand (DASH) | 3 mo, 6 mo, 1 year, 2 years
Quality of life assessed with 15D | 6 weeks, 3 mo, 6 mo, 1 year, 2 years
Subjective satisfaction | 6 weeks, 3 mo, 6 mo, 1 year, 2 years
Complications | 6 weeks, 3 mo, 6 mo, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Lähdeoja, MD, Principal Investigator — University of Helsinki; Mika Paavola, MD, PhD, Study Director — University of Helsinki; Jarkko Pajarinen, MD, PhD, Study Director — University of Helsinki; Seppo Koskinen, MD, PhD, Study Chair — University of Helsinki
Locations (1):
- Töölö Hospital Trauma Center, Helsinki University Central Hospital,, Helsinki, Finland

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196